CLINICAL TRIAL: NCT03302832
Title: Effectiveness of Reduced Frequency Physical Therapy Supplemented With In-home Exercise Equipment Compared to Standard Care Physical Therapy in Total Knee Arthroplasty
Brief Title: Effectiveness of Reduced Frequency Physical Therapy in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campbell University, Incorporated (Other)
Responsible Party: Principal Investigator, Bradley Myers, Assistant Professor, Campbell University, Incorporated
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 313
Record Dates: First submitted 2017-09-22; First posted 2017-10-05 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Knee Osteoarthritis; Knee Arthritis; Knee Arthropathy
Keywords: Total Knee Arthroplasty; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Physical Therapy (Active Comparator): The participants randomized to the Standard Care Physical Therapy group will begin outpatient physical therapy services after discharge from inpatient care, on day 4 or 5 post-Total Knee Arthroplasty. The frequency of sessions will be 2-3 x per week for the initial 2 weeks, followed by 2 x per week until the culmination of physical therapy. The frequency and duration of sessions will be determined by the treating physical therapist based upon the clinical needs and progress of the specific participant.
  Interventions: Other: Physical Therapy
- Physical Therapy and in-Home Equipment (Experimental): The participants randomized to the experimental group will begin outpatient physical therapy services after discharge from inpatient care, on day 4 or 5 post-Total Knee Arthroplasty. The frequency of physical therapy sessions will be 1 x per week throughout the duration of the study period. In addition, this group will utilize in-home exercise equipment daily.
  Interventions: Other: Physical Therapy; Other: In-home Exercise Equipment

INTERVENTIONS:
Other: Physical Therapy — Physical therapy includes both the in-person and home-based interventions prescribed for each individual participant in order to maximize overall patient outcomes including: ambulation, range of motion, strength, functional activities, pain, swelling, balance, patient safety, and other items within the scope of physical therapy practice.
Other: In-home Exercise Equipment — The in-home exercise component of the study will supplement physical therapy services. This exercise equipment will be utilized daily for up to 90 minutes as guided by the healthcare team
  Other Names: Total Range Exerciser Arc; T-REX Arc
  Arms: Physical Therapy and in-Home Equipment

SUMMARY:
Rehabilitation after Total Knee Arthroplasty surgery involves physical therapy services to address limitations in range of motion, strength, and participation in normal daily activities. This investigation will compare the outcomes from standard physical therapy intervention in comparison to reduced frequency physical therapy sessions supplemented with in-home exercise equipment.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a common surgical procedure for individuals experiencing pain and reduced physical abilities related to knee pain, most commonly osteoarthritis. Common physical impairments associated with post-operative TKA rehabilitation include: reduced knee range of motion (ROM), reduced strength, reduced participation in activities of daily living, and pain. TKA surgery is routinely paired with physical therapy (PT) interventions post-operatively in order to facilitate recovery for patients electing to undergo this intervention. The Total Range Exerciser (T-REX) is a medical device aimed at reducing the need for post-operative physical therapy services while promoting outcomes.

A successful outcome after total knee arthroplasty requires symptom relief and restoration of physical function. Measurement of pain and function can be achieved through patient-reported outcomes measures and objective functional testing. The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a patient-reported outcomes measure intended to capture the individual patient's perception of progress throughout the rehabilitative process. Objective measurements of physical function are necessary to quantify the magnitude of physical impairment associated with the patient's perceived status. Physical function can be measured through standardized assessment of knee ROM, strength, and ambulation. The purpose of this study is to evaluate the effectiveness of standard physical therapy compared to reduced frequency physical therapy supplemented with the (T-REX) after in total knee arthroplasty in subjective and objective measurements of physical function.

ELIGIBILITY:
Inclusion Criteria:

* Individual is to undergo TKA by a licensed physician at Participating hospital group
* Participating primary health insurance provider
* Patient is < 64.5 years of age
* Willingness to participate in study protocol

Exclusion Criteria:

* Previous or current history of cancer
* High risk for cardiovascular disease as determined by the American College of Sports Medicine
* Individuals with documented mental, psychiatric, or emotional disabilities
* Inability to read and write in English

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) | Pre-surgery to 3 months post-surgery
  The KOOS measurement is a patient-reported questionnaire that contains 42 questions covering 5 categories (pain, symptoms, activities of daily living, sports and recreation, and quality of life

SECONDARY OUTCOMES:
Self-reported home exercise compliance/adherence | 1 month post-surgery, 2 months post-surgery, 3 months post-surgery
  Basic questions regarding the percent compliance with home exercises, amount of exercise time per week, and amount of days the participant performed exercise each week.
Change in Knee Active Range of Motion (AROM) | Pre-surgery to 3 months post-surgery
  Measurement of the range of motion that the participant can perform (in degrees) when maximally bending and straightening the knee.
Change in Knee Passive Range of Motion (PROM) | Pre-surgery to 3 months post-surgery
  Measurement of the range of motion (in degrees) that the participant's knee can maximally bend and straighten as a result of a manually applied movement.
Change in Timed Up-and-Go Test (TUG) | Pre-surgery to 3 months post-surgery
  The TUG is a physical performance test that consists of the participant rising from a chair, ambulating 9 meters, turning around, returning to the chair and sitting. It is recorded in seconds.
Change in 6-minute Walk Test (6MWT) | Pre-surgery to 3 months post-surgery
  The 6MWT is an assessment of longer duration ambulation and cardiorespiratory endurance. The test measurement is the total amount of distance that the participant ambulates within a 6-minute period.
Change in 30 second Chair Stand Test (30s-CST) | Pre-surgery to 3 months post-surgery
  The 30s-CST is a test of strength, endurance and functional balance. The maximum number of sit to stand repetitions performed over a 30 second period represents the score for this test. Pre-test positioning includes placement of a 44 cm (17 inch) chair, measured from floor to seat surface, against a wall to inhibit movement of the chair during the test.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Myers, PT, DPT, DSc, Principal Investigator — Assistant Professor
Locations (1):
- EmergeOrtho, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No data is intended to be shared with other researchers